CLINICAL TRIAL: NCT00944775
Title: Effects of Exercise Training on Non-invasive Cardiac Measures in Patients Undergoing Long-term Hemodialysis: A Randomized Controlled Trial
Brief Title: Exercise and Cardiac Measures in Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Evangelia Kouidi, Professor of Sports Medicine, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: RenalRehab
Record Dates: First submitted 2009-04-09; First posted 2009-07-23 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Sudden Cardiac Death
Keywords: Exercise; Dialysis; Non-invasive cardiac measures; Exercise trained patients; Controls
MeSH Terms: conditions — Death, Sudden, Cardiac; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- exercise training (Experimental): 10-month exercise training program
  Interventions: Behavioral: Exercise training
- controls (No Intervention): usual care sedentary lifestyle

INTERVENTIONS:
Behavioral: Exercise training — 10-month exercise training program during hemodialysis sessions
  Other Names: Group A; group B
  Arms: exercise training

SUMMARY:
Background: The impact of the known non-invasive cardiac indices for identification of hemodialysis (HD) patients at high-risk for sudden cardiac death (SCD) has not been evaluated.

Patients: Fifty-nine HD patients were randomized into 2 groups. Thirty of them (group A-aged 54.6±8.9 years) participated in a supervised training program with stationary bicycles during their HD sessions (3/weekly) for 10 months, while the rest (group B-aged 53.2±6.1 years) remained untrained and were used as controls.

Study hypothesis: Exercise training will affect most of the non-invasive cardiac markers of SCD and the total score positively.

Method: At entry, as well as at the end of the study all subjects underwent a cardiopulmonary exercise testing (estimation of aerobic capacity-VO2peak), an echocardiographic study (LV ejection fraction -LVEF evaluation), an ambulatory 24-hour Holter monitoring for cardiac autonomic nervous system activity evaluation by time- and frequency- domain heart rate variability (HRV) calculation (measurement of SDNN, mean RR and low to high frequency ratio-LF/HF), a signal-averaged ECG (late potentials-LP documentation) and a submaximal exercise test for microvolt-T-wave alternans (TWA) detection.

DETAILED DESCRIPTION:
The identification of patients on hemodialysis (HD) at increased cardiac risk with powerful screening tests and the reduction of factors, which increase the probability of malignant arrhythmias are important for primary prevention of sudden cardiac death (SCD).

Study Design: randomized and controlled clinical trial. Setting & Participants: Fifty-nine HD patients were randomized into exercise training group (group A-30 patients) and controls (group B-29 patients).

Intervention: Group A participated in a 10-month supervised exercise training program during the HD sessions (3/weekly).

Outcomes: The effects of exercise on the score of the non-invasive cardiac markers for SCD risk stratification and on the occurrence of each variable separately. Statistical analysis included a two-group comparison of change scores and an analysis of covariance adjusting for baseline.

Measurements: At entry and the end of the study, in all participants aerobic capacity (VO2peak) and left ventricular ejection fraction (LVEF) were estimated, late potentials and T-wave alternans were detected and heart rate variability was calculated. Specifically, from the 24-h Holter monitoring the standard deviation of all the normal R-R intervals (SDNN), the mean R-R intervals (mean RR), the low (LF) and high (HF) frequency components of the autoregressive power spectrum of the NN intervals and their ratio (LF/HF) were recorded.

ELIGIBILITY:
Inclusion Criteria:

* on HD for at least 6 months
* in sinus rhythm
* able to reach a sufficient workload during ergometry

Exclusion Criteria:

* with bundle branch block
* unstable hypertension
* diabetes mellitus
* severe congestive heart failure
* recent myocardial infarction
* unstable angina

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2007-08; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The composite risk score | at entry and after 10 months

SECONDARY OUTCOMES:
aerobic capacity (VO2peak) | At entry and after 10 months
Left ventricular ejection fraction (EF)- echocardiography | At entry and after 10 months
standard deviation of normal R-R intervals- SDNN (holter monitoring) | At entry and after 10 months
positive T-wave alternans and Late potentials | At entry and after 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Evangelia J Kouidi, Associate Pr, Principal Investigator — Aristotle University of Thessaloniki, Greece
Locations (1):
- Laboratory of Sports Medicine, Thessaloniki, Greece

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639
- [Derived] Kouidi EJ, Grekas DM, Deligiannis AP. Effects of exercise training on noninvasive cardiac measures in patients undergoing long-term hemodialysis: a randomized controlled trial. Am J Kidney Dis. 2009 Sep;54(3):511-21. doi: 10.1053/j.ajkd.2009.03.009. Epub 2009 Jul 30. PMID 19646801